CLINICAL TRIAL: NCT00493311
Title: A Phase III, Randomized, Double-Blind, Placebo-Controlled, Single-Dose Study of the Efficacy and Safety of Intravenous Acetaminophen Versus Placebo for the Treatment of Endotoxin-Induced Fever in Healthy Adult Males
Brief Title: Safety of Intravenous Acetaminophen Vs Placebo for the Treatment of Endotoxin-Induced Fever in Healthy Adult Males
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CPI-APF-302
Record Dates: First submitted 2007-06-27; First posted 2007-06-28 (Estimated); Results first posted 2010-09-21 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-10

CONDITIONS: Fever
MeSH Terms: conditions — Fever | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- IV Acetaminophen (Experimental): 1 g of acetaminophen in 100 mL of intravenous solution
  Interventions: Drug: IV Acetaminophen; Biological: Reference Standard Endotoxin (RSE)
- IV Placebo (Placebo Comparator): 100 mL of intravenous placebo solution
  Interventions: Drug: IV Placebo; Biological: Reference Standard Endotoxin (RSE)

INTERVENTIONS:
Drug: IV Placebo — IV Placebo
  Other Names: Placebo
  Arms: IV Placebo
Drug: IV Acetaminophen — Intravenous acetaminophen solution 1 g / 100 ml
  Other Names: IV APAP; APAP
  Arms: IV Acetaminophen
Biological: Reference Standard Endotoxin (RSE) — Administration of Reference Standard Endotoxin (RSE) to induce fever. Applicable to both study arms: Administration of a 1 ng/kg body weight test dose of RSE to test for fever response. Observation period of at least 60 minutes to ensure no exaggerated systemic responses, followed by administration of a 4 ng/kg of RSE to induce fever.
  Other Names: IV Acetaminophen; APAP

SUMMARY:
A research study to determine if acetaminophen (APAP) given intravenously (IV-a liquid given through a needle into a vein in your arm) is safe and effective in controlling fever when compared to placebo. Acetaminophen given this way is the investigational part of this study.

DETAILED DESCRIPTION:
A Phase III, Randomized, Double-Blind, Placebo-Controlled, Single-Dose Study of the Efficacy and Safety of Intravenous Acetaminophen (IVAPAP) Versus Placebo for the Treatment of Endotoxin-Induced Fever in Healthy Adult Males

ELIGIBILITY:
Inclusion Criteria:

* Provide written Informed Consent prior to participation in the Study
* Be a healthy male between the ages of 18 and 75 years of age, inclusive, at Randomization
* Have a Body Mass Index (BMI) ≥ 19 and ≤ 40 lbs / in2
* Have the ability to read and understand the Study procedures and have the ability to communicate meaningfully with the Study Investigator and staff
* Be free of physical, mental, or medical conditions which, in the opinion of the Investigator, may confound quantifying assessments for the Study
* Be willing to abstain from smoking cigarettes or using nicotine products from the time of admission to Clinic until Study Completion

Inclusion Criteria (Pre-Randomization) To be eligible for entry into the Study, Subjects must meet each of the following criteria prior to Randomization:

* Be free of evidence of infection based upon clinical assessment and blood (Complete Blood Count-CBC) and urine testing
* Have an average baseline oral temperature that is equal to or below 37 ºC (98.6 ºF) and does not vary more than 0.4 ºC (0.7 ºF) from lowest to highest on three assessments performed during a 30 minute period
* Not develop a medically significant allergic or exaggerated systemic response to administration of a test dose of reference standard endotoxin
* Develop a core temperature of at least 38.6 ºC (101.5 ºF) after intravenous reference standard endotoxin dosed per Study guidelines and have a fever response to endotoxin that is at or near the peak temperature by virtue of two consecutive temperature assessments 5 minutes apart that are within 0.2 ºC (0.4 ºF) of each other

Exclusion Criteria:

* Has been treated with any medication having antipyretic effects (e.g., corticosteroid, Non-steroidal anti-inflammatory drug (NSAID), aspirin or acetaminophen) within 2 days of clinic admission (aspirin at low dose for cardiac prophylaxis is allowed, but should not be taken on the day of the Study)
* Has significant medical disease(s), laboratory abnormalities, or condition(s) that in the Investigator's judgment could compromise the Subject's welfare, ability to communicate with the Study staff, complete Study activities, or would otherwise contraindicate Study participation.
* Has known hypersensitivity or contraindication to receiving endotoxin that in the Investigator's clinical judgment merits discontinuation from further Study participation
* Has known hypersensitivity to acetaminophen, the inactive ingredients (excipients) of the Intravenous(IV) acetaminophen formulation or the Rescue Medications (ibuprofen, aspirin and ketorolac)
* Has known or suspected recent history of alcohol or drug abuse or dependence as defined by Diagnostic and Statistical Manual of Mental Disorders, 4th Edition (DSM-IV) criteria
* Has a history of nasal polyps, angioedema, significant or actively treated bronchospastic disease, or any other significant medical condition that contraindicates participation in the Study or receiving endotoxin, Study Medication, or Rescue Medication
* Has an active infection or other disease or condition that may cause abnormal alterations in body temperature, or has worked the night shift on a regular basis for the last 3 months prior to Screening
* Has impaired liver function, e.g. Alanine aminotransferases (ALT) greater than or equal to 3 times the upper limit of normal, bilirubin greater than 3.0, active hepatic disease, or evidence of clinically significant liver disease (e.g., cirrhosis or hepatitis)
* Has participated in another clinical Study (investigational or marketed product) within 30 days of Screening

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-06; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Scirex Research Center, Austin, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited at a single clinical research facility in the United States during July to September 2007.
Pre-assignment Details: Eligible subjects received intravenous endotoxin to induce fever and were then randomized to receive either 1 g acetaminophen in 100 ml intravenous solution or 100 ml placebo solution.
Groups:
- Intravenous (IV) Placebo: After induction of fever by endotoxin administration, subjects received one infusion of 100 ml intravenous placebo solution
- Intravenous (IV) Acetaminophen 1 g: After induction of fever by endotoxin administration, subjects received one infusion of 1 g of acetaminophen in 100 ml intravenous solution
Period: Overall Study
Arm/Group | Intravenous (IV) Placebo | Intravenous (IV) Acetaminophen 1 g
Started | 29 | 31
Completed | 27 | 29
Not Completed | 2 | 2
Not completed — Need for rescue medication | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intravenous (IV) Placebo | Intravenous (IV) Acetaminophen 1 g | Total
Number analyzed (Participants) | 29 | 31 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 31 | 60
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.0 (10.02) | 29.7 (7.35) | 29.9 (8.67)
Sex: Female, Male [Count of Participants; unit: Participants] — Only male subjects were allowed to participate in the study.
  Participants
    Female | 0 | 0 | 0
    Male | 29 | 31 | 60
Region of Enrollment [Number; unit: participants]
  United States | 29 | 31 | 60

OUTCOME MEASURES:

1. Primary Outcome: Weighted Sum of Temperature Differences Over 6 Hours (WSTD6) Assessment of the Antipyretic Effect Over 6 h of a Single Dose of IV APAP vs. Placebo for Treatment of Endotoxin-induced Fever
Description: The primary efficacy endpoint was WSTD6 defined as the weighted sum of temperature differences from the temperature at each assessment timepoint through 6 hours compared with the temperature at T0, weighted by the time elapsed between each 2 consecutive timepoints.
Time Frame: Baseline (T0) to 6 hours post study drug administration
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | Intravenous (IV) Placebo | Intravenous (IV) Acetaminophen 1 g
Number analyzed (Participants) | 29 | 31
Degrees Celsius | -0.7 (3.32) | -3.7 (3.58)

2. Secondary Outcome: Weighted Sum of Temperature Differences Over 3 Hours (WSTD3) Assessment of the Antipyretic Effect Over 3 Hours of a Single Dose of IV APAP vs. Placebo for Treatment of Endotoxin-induced Fever.
Description: WSTD3 is defined as the weighted sum of temperature differences from the temperature at each assessment timepoint through the first 3 hours compared with the temperature at T0, weighted by the time elapsed between each 2 consecutive timepoints.
Time Frame: Baseline (T0) to 3 hours
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | Intravenous (IV) Placebo | Intravenous (IV) Acetaminophen 1 g
Number analyzed (Participants) | 29 | 31
Degrees Celsius | 0.7 (1.36) | -0.9 (1.35)

3. Secondary Outcome: Maximum Temperature Change During the Period From T0 to T360 Minutes (6 Hours After Study Drug Administration)
Time Frame: Baseline (T0) to 360 minutes (6 hours) post study drug administration
Measure: Mean (Standard Deviation); unit: Degrees celsius
Arm/Group | Intravenous (IV) Placebo | Intravenous (IV) Acetaminophen 1 g
Number analyzed (Participants) | 29 | 31
Degrees celsius | -0.9 (0.75) | -1.3 (0.65)

4. Secondary Outcome: The Percentage of Subjects With Temperature Less Than 38 Degrees Celsius at Any Timepoint During the Time From T0 to T360 Minutes (6 Hours After Study Drug Administration)
Time Frame: 360 minutes (6 hours after study drug administration)
Measure: Number; unit: Percentage of participants
Arm/Group | Intravenous (IV) Placebo | Intravenous (IV) Acetaminophen 1 g
Number analyzed (Participants) | 29 | 31
Percentage of participants | 3 | 13

5. Secondary Outcome: Global Assessment of Treatment at T360 Minutes or Early Termination.
Description: Subject Global Evaluation was assessed by subject using a 4 point categorical scale in response to the following question:Overall, how would you rate the study treatments? 0 = Poor
  1. = Fair
  2. = Good
  3. = Excellent
Time Frame: Baseline (T0) to 6 hours
Measure: Number; unit: participants
Arm/Group | Intravenous (IV) Placebo | Intravenous (IV) Acetaminophen 1 g
Number analyzed (Participants) | 29 | 31
participants
  Rate treatment as 'poor' | 2 | 1
  Rate treatment as 'fair' | 9 | 5
  Rate treatment as 'good' | 10 | 16
  Rate treatment as 'excellent' | 8 | 9

ADVERSE EVENTS:
Time Frame: Treatment Emergent Adverse Events(TEAEs)were reported from T0 (on or after the start of study medication) to 6 hours after study medication was administered to the subject.
Description: TEAEs are adverse events that start on or after the study medication is given to the subject.
Arm/Group | Intravenous (IV) Placebo | Intravenous (IV) Acetaminophen 1 g
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/31
Other Adverse Events (participants affected / at risk) | 13/29 | 14/31
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Intravenous (IV) Placebo (N=29) | Intravenous (IV) Acetaminophen 1 g (N=31)
Alanine aminotransferase increased (Investigations) | 6 | 5
Aspartate aminotransferase increased (Investigations) | 4 | 6
Blood bilirubin increased (Investigations) | 1 | 3
Diarrhoea (Gastrointestinal disorders) | 3 | 1
Dizziness (Nervous system disorders) | 2 | 2
Gamma-glutamyltransferase increased (Investigations) | 8 | 5
Mucosal dryness (General disorders) | 2 | 1
Nausea (Gastrointestinal disorders) | 4 | 2
Vomiting (Gastrointestinal disorders) | 3 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 1
Headache (Nervous system disorders) | 3 | 0
Somnolence (Nervous system disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator may publish only after cooperative publication or 18 months after sponsor's final evaluation of study data, whichever occurs first. At least 60 days prior to submission for publication, investigator must submit manuscript to sponsor for review and comment. Sponsor has 60 day period thereafter to respond with comment. Investigator will remove confidential information at the request of sponsor.